CLINICAL TRIAL: NCT00791973
Title: Effect of Veramyst on the Nasal and Ocular Symptoms of the Early Reaction to Nasal Challenge With Allergen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, MD, University of Chicago
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 16367B (OC 3)
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Veramyst, then Placebo (Active Comparator): fluticasone furoate (Veramyst) nasal spray once daily for a week, then one week washout period followed by placebo nasal spray once daily for a week
  Interventions: Drug: fluticasone furoate; Drug: Placebo
- Placebo, then Veramyst (Active Comparator): placebo nasal spray once daily for a week, then one week washout period followed by fluticasone furoate (veramyst) nasal spray once daily for a week
  Interventions: Drug: fluticasone furoate; Drug: Placebo

INTERVENTIONS:
Drug: fluticasone furoate — 2 puffs in each nostril once daily for 1 week
  Other Names: Veramyst
Drug: Placebo — 2 puffs in each nostril once daily for 1 week

SUMMARY:
The purpose of this study is to help us to a better understanding of how nose and eye symptoms are related in patients with allergies.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 45 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 subjects were screened for eligibility
Pre-assignment Details: 15 of the 24 subjects screened were eligible for the study and were randomly assigned to groups
Groups:
- Veramyst, Then Placebo: fluticasone furoate (Veramyst) nasal spray once daily, 2 puffs/nostril, for a week, then one week washout period followed by placebo nasal spray once daily , 2 puffs/nostril, for a week
- Placebo, Then Veramyst: placebo nasal spray once daily (2 puffs/nostril) for a week, then one week washout period followed by fluticasone furoate (veramyst) nasal spray once daily (2 puffs/nostril) for a week
Period: First Intervention (1 Week)
Arm/Group | Veramyst, Then Placebo | Placebo, Then Veramyst
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Veramyst, Then Placebo | Placebo, Then Veramyst
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Veramyst, Then Placebo | Placebo, Then Veramyst
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Veramyst, Then Placbeo: fluticasone furoate (Veramyst) nasal spray once daily, 2 puffs/nostril, for a week, then one week washout period followed by placebo nasal spray once daily , 2 puffs/nostril, for a week
- Total: Total of all reporting groups
Arm/Group | Veramyst, Then Placbeo | Placebo, Then Veramyst | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11) | 29 (6) | 30 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Tryptase Level From Baseline to Post-antigen Challenge
Description: Tryptase levels (mcg/L) were measured from nasal lavages
Time Frame: After one week of treatment wtih veramyst or placebo
Measure: Median (Inter-Quartile Range); unit: mcg/L
Groups:
- Veramyst: fluticasone furoate (Veramyst) nasal spray once daily, 2 puffs/nostril, for a week
- Placebo: placebo nasal spray once daily (2 puffs/nostril) for a week
Arm/Group | Veramyst | Placebo
Number analyzed (Participants) | 15 | 15
mcg/L | 0 [0 to 11.8] | 2.31 [0 to 8.8]
Statistical Analysis 1: Comparison: Veramyst vs Placebo; Test type: Superiority or Other; p = 0.33, Wilcoxon signed-rank test

2. Secondary Outcome: Total Eye Symptom Scores After Antigen Challenge
Description: Watery and itchy eye symptoms will be scored based on the following scale: 0=no symptoms, 1= mild, 2= moderate, 3= severe
Time Frame: After one week of treatment wtih veramyst or placebo
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Veramyst | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 3 [0 to 4] | 3 [1 to 9]
Statistical Analysis 1: Comparison: Veramyst vs Placebo; Test type: Superiority or Other; p = 0.14, Wilcoxon signed-rank test

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Veramyst | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes